CLINICAL TRIAL: NCT03327415
Title: The French National Survey on Food Consumption of Children Under 3 Years of Age
Brief Title: Nutri-Bébé 2013 Survey on Food Consumption of Infants and Young Children
Acronym: NBB2013
Status: Completed | Type: Observational
Sponsor: Secteur Français des Aliments de l'Enfance (Industry)
Collaborators: TNS Sofres polling institute (Unknown); Centre de Recherche pour l'Etude et l'Observation des Conditions de Vie (Unknown)
Responsible Party: Sponsor
Other Study IDs: Nutri-Bébé SFAE 2013
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Food Consumption; Infants; Toddlers
Keywords: Children; Food practice; Food consumption; Nutrient intake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Age groups: Eleven age groups that took into account the previous surveys and the key stages of child development were defined: 15 days to 3 months, 4, 5, 6, 7, 8-9, 10-11, 12- 17, 18-23, 24-29, and 30-35 months.

SUMMARY:
The Nutri-Bébé 2013 survey is an observational cross-sectional study aiming to update food consumption, practices and nutrient intakes in children under 3 years of age in metropolitan France.

DETAILED DESCRIPTION:
Nutri-Bébé 2013 is the 5th edition of a survey conducted every 8 years since 1981 by the SFAE. The Nutri-Bébé 2013 survey is an observational cross-sectional study conducted in children living in France aged 15 days to 35 months by an official polling institute, the TNS Sofres according to the guidelines laid down in the Declaration of Helsinki. TNS Sofres fulfills the following standards and industry requirements (ESOMAR professional code of conduct and standards, ISO 20252:2012 international standard for market, opinion and social research, French data protection act (loi "informatique et libertés "). TNS Sofres ensures to conduct the surveys in accordance with the regulation on personal data protection and that respondents' personal identity is withheld. Moreover TNS Sofres appointed a data protection officer, the "Correspondant Informatique et Libertés", who is the point of contact between the "Commission Nationale de l'Informatique et des Libertés" (CNIL), the French data protection authority) and the company. The company is thus exempted, of the notification process to the CNIL. Given the type of survey conducted, namely a survey of consumption, and the characteristics developed above, the study does not require any opinion of the ethics committee.

The survey includes a section on eating behaviours and a section on food consumption.

After giving their informed consent, parents had to record the food consumption during 3 non-consecutive days (2 week days and one weekend day)framed by two face-to-face interviews,. A second visit occurred seven days later to verify and complete the diary if necessary, and conduct a face-to-face interview with the mother about eating habits over the survey period. Both interviews were recorded using CAPI® software (Computer Assisted Personal Interviews, http://www.soft-concept.com). During this visit, the child was weighed (naked, with a clean diaper or underwear) using a Tefal PREMISS PP1000VO scale with a precision of 100 g.

The child's food consumption diary was completed between the two visits of the TNS Sofres investigator. The person in charge of the child was trained to qualitatively and quantitatively report all liquid and solid foods consumed and all drinks, by specifying the exact name of the product, its potential trademark or whether it was "homemade". The type of water consumed was noted as being either "bottled" or "tap". The type (breakfast, morning snack, lunch, afternoon snack, dinner, nocturnal food intake) and timing of food consumption were collected. If applicable, vitamin, mineral or medicine supplements were noted. During the second visit the investigator reviewed thoroughly the record with the caregiver and checked the way of reporting the quantities as well as the interpretation of the photographic tool kit in order to be as close as possible to reality.

ELIGIBILITY:
Inclusion Criteria:

* informed parental consent to participate in the study,
* absence of intercurrent or chronic disease
* birth weight above 2.5 kg

Exclusion Criteria:

* Non compliance withe the study protocol
* For outcome 3 analysis (intakes), reported weight inconsistent with the child's age (> or <3 SD)

Age Groups: Child, Adult, Older Adult
Study Population: The present survey is based on a randomly selected sample with socio-demographic characteristics similar to the general population living in mainland France (i.e. excluding Corsica, overseas departments, regions, and communities, and New Caledonia). A quota sampling method was used: sampling wastratified by residential area, size of the urban agglomeration, infant gender, mother's professional activity, occupational and socio-occupational status and adjusted for these different characteristics. This stratification was based on the population characteristics of the 2002 census of the National Institute for Statistics and Economic Research (INSEE, Institut National de la Statistique et des Etudes Economiques).
Sampling Method: Probability Sample
Enrollment: 1192 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2013-04-21 (Actual); Study Completion 2015-02-15 (Actual)

PRIMARY OUTCOMES:
Age at inclusion | January to april 2013
  months
Weight at inclusion | January to april 2013
  kg
Prevalence of socio-demographic condition, feeding practice, consumption energy contribution, | January to april 2013
  frequency in %
Time of introducing or withdrawing a food | history of feeding before being included in the survey
  months
Mean over 3 days of Food quantities and macronutrient intake (water, protein, lipid, carbohydrate, fiber) | January to april 2013
  g/d
Mean over 3 days of Intakes of Linoleic-, alpha linolenic-acids, DHA, ARA, minerals (sodiu, calcium, phosphorus, magnesium, iron, zinc), Vitamin B1,B2, B3, B6, C, E | January to april 2013
  mg/d
Mean over 3 days of intakes of Vitamin B9, B12, Retinol, Beta-caroten | January to april 2013
  micro g/d
Vitamin A intake | January to april 2013
  RE(Retinol Equivalent)/d

SECONDARY OUTCOMES:
Nutrient intakes per kilogram body weight | January to april 2013
  unit/kg/d
Comparison with 2005 data | 2013 vs 2005
  p value

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel TAVOULARIS, Engineer,MSc, Principal Investigator — CREDOC; Yves EMERY, MSc, Principal Investigator — TNS Sofres; Jean-Pierre CHOURAQUI, MD, MSc, Principal Investigator — CHUV Lausanne; Magali BOCQUET, Engineer,MSc, Study Director — Secteur Français des Aliments de l'Enfance
Locations (1):
- EMERY Yves, Montrouge, France

IPD SHARING:
Plan to Share IPD: No
To be shared is the global report of results on each items (food practices, food consumption, nutrients intakes), according to age groups.

REFERENCES:
- [Derived] Chouraqui JP, Renella R, Turck D. Assessment of Dietary Iron Intake and Sources in Early Childhood in a Nationally Representative Cross-Sectional Survey. J Acad Nutr Diet. 2024 Jul;124(7):823-832.e1. doi: 10.1016/j.jand.2023.12.009. Epub 2023 Dec 22. PMID 38142742
- [Derived] Chouraqui JP, Darmaun D, Salmon-Legagneur A, Shamir R. Protein intake pattern in non-breastfed infants and toddlers: A survey in a nationally representative sample of French children. Clin Nutr. 2022 Feb;41(2):269-278. doi: 10.1016/j.clnu.2021.12.006. Epub 2021 Dec 8. PMID 34998033